CLINICAL TRIAL: NCT03191136
Title: A Open-label, Randomized, Single Dose, Crossover Clinical Trial to Assess the Effect of Food on the Pharmacokinetics of YHD1119 in Healthy Male Volunteers
Brief Title: Clinical Trial to Assess the Effect of Food on the Pharmacokinetics of YHD1119 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHD1119-104
Record Dates: First submitted 2017-05-24; First posted 2017-06-19 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2017-06

CONDITIONS: Peripheral Neuropathic Pain

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, single dose, cross-over clincial trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental): taking YHD1119 (pregabalin 300mg) in fasted state at Period 1
  Interventions: Drug: YHD1119 300mg
- Group2 (Experimental): taking YHD1119 (pregabalin 300mg) in fed state at Period 1
  Interventions: Drug: YHD1119 300mg

INTERVENTIONS:
Drug: YHD1119 300mg — Period 1:a single dose of YHD1119 300mg is administered in fasting condition Period 2:a single dose of YHD1119 300mg is administered in fed condition
Drug: YHD1119 300mg — Period 1:a single dose of YHD1119 300mg is administered in fed condition Period 2:a single dose of YHD1119 300mg is administered in fasting condition

SUMMARY:
This is a phase 1, open-label, randomized, single dose, crossover clinical trial to assess the effect of food on the pharmacokinetics of YHD1119 in healthy male volunteers.

Hypothesis: "YHD1119" is showing equal equal pharmacokinetics in fasted and fed state.

DETAILED DESCRIPTION:
This is a phase 1, open-label, randomized, single dose, crossover clinical trial to assess the effect of food on the pharmacokinetics of YHD1119 in healthy male volunteers.

Group 1: 12 subjects will be assigned and they will be administered YHD1119 in fasted state at Day 1 and in fed state at Day 8.

Group 2: 12 subjects will be assigned and they will be administered YHD1119 in fed state at Day 1 and in fasted state at Day 8.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male with body mass index(BMI) between 18.5 and 30 kg/m2
* Who has not suffered from clinically significant disease
* Provision of signed written informed consent

Exclusion Criteria:

* History of and clinically significant disease
* A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs
* Administration of other investigational products within 3 months prior to the first dosing
* Volunteers considered not eligible for the clinical trial by the investigator due to reasons including laboratory test results, ECGs, or vital signs

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male with body mass index (BMI) between 18.5kg/m2 and 30kg/m2
Enrollment: 24 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
YHD1119 Cmax | 0 - 36hrs
  Cmax
YHD1119 AUC last | 0 - 36hrs
  AUC last

CONTACTS AND LOCATIONS:
Overall Officials: Mingul Kim, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moon SJ, Jeon JY, Lim Y, An T, Jang SB, Kim S, Na WS, Lee SY, Kim MG. Pharmacokinetics of a New, Once-Daily, Sustained-release Pregabalin Tablet in Healthy Male Volunteers. Clin Ther. 2021 Aug;43(8):1381-1391.e1. doi: 10.1016/j.clinthera.2021.06.010. Epub 2021 Jul 11. PMID 34256964